CLINICAL TRIAL: NCT04811170
Title: The Effectiveness of Counselling on Mood Symptoms of Low-income Ethnic Minorities in Hong Kong: a Wait-list Randomised Controlled Trial
Brief Title: Counselling Service for Low-income EM in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Zubin Foundation (Unknown)
Responsible Party: Principal Investigator, Professor Eric Y.H. Chen, Chair Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EM RCT
Record Dates: First submitted 2021-03-06; First posted 2021-03-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Counselling group (Experimental): Counselling sessions will be conducted at the designated centers operated by the Zubin foundation. According to the level of the DASS score, 6 to 10 sessions (based on the algorithm) of counselling service will be provided to the participants by three registered counsellors. A lead counsellor will oversee all cases and services. The counselling program consists of 6-10 60-minute sessions, and the sessions can be flexibly delivered over 1 to 2 weeks, ranging from one 60-minute session biweekly or weekly.
  Interventions: Other: Counselling
- Waiting group (Other): For participants in the waiting list control group, they will receive monitoring service over phone calls during the 8-12 weeks wait period. Counselling service will be offered after the post-treatment assessment.
  Interventions: Other: Counselling

INTERVENTIONS:
Other: Counselling — Participants with mild to moderate mood symptoms will receive a maximum of 6 counselling sessions and will be assessed at baseline (T0, W1), at post-treatment for counselling group (T1, W8), and after 2 booster sessions. Participants in the waiting list control group will receive the same counselling service after the counselling group completed the intervention. Participants with severe mood symptoms will receive a maximum of 10 counselling sessions and will be assessed at baseline (T0, W1), at post-treatment for counselling group (T1, W12), and after 2 booster sessions. Participants in the waiting list control group will receive the same counselling service after the counselling group completed the intervention.

SUMMARY:
This study will recruit 120 ethnic minorities in Hong Kong from the Zubin Foundation (TZF) at the Ethnic Minority Well-being Centre (EMWBC), which is a service provider of EM mental health support in Hong Kong. This service provides counselling service and referrals to HA via the Integrated Community Centre for Mental Wellness (ICCMW) to psychiatrists. The service covers the South Asians population of approximately eighty-four thousands people in Hong Kong. Participants will be recruited by the Zubin Foundation through outreach activities screening and counselling will be conducted in partnering schools and NGOs (e.g., Yan Oi Tong in Tuen Mun and Yew Chung College of Early Childhood Education in Aberdeen).

The study aims to evaluate the effectiveness of counselling service for improving mood symptoms in EM, also to assess the effectiveness of counselling service in improving psychological functioning (i.e. resilience and rumination, self-compassion, self-efficacy and life satisfaction), social functioning and quality of life and to assess whether the counselling service is cost-effective and offers good value for money.

The study is a wait-list RCT. Participants will be randomly assigned into either the intervention group (n = 60) or the wait-list control group (n = 60) in a 1:1 ratio. Each participant in the intervention group will be paired up with a participant from the control group, the number of sessions and duration of waiting period varies depending on the severity of mood symptoms. Participants with mild to moderate mood symptoms will receive a maximum of 6 counselling sessions and will be assessed at baseline (T0, W1), at post

-treatment for counselling group (T1, W8), and after 2 booster sessions. Participants in the waiting list control group will receive the same counselling service after the counselling group completed the intervention. Participants with severe mood symptoms will receive a maximum of 10 counselling sessions and will be assessed at baseline (T0, W1), at post-treatment for counselling group (T1, W12), and after 2 booster sessions. Participants in the waiting list control group will receive the same counselling service after the counselling group completed the intervention.

This evaluation study will provide data to inform the government in mental health policy review and development.

ELIGIBILITY:
Inclusion Criteria:

* South Asian ethnic minorities (except domestic helper) in Hong Kong;
* 15 - 64 years
* reach at least the mild level of the Depression Anxiety Stress Scales - 21 Items in at least one of the following scores: the Depression Score (DASS-D), Anxiety Score (DASS-A) or Stress Score (DASS-S), or low Quality of Life score
* have sufficient proficiency in English, Hindi or Urdu to understand verbal instructions and give informed consent.

Exclusion Criteria:

* from high-income family (cut off ranges from HK$15K for single person family to HK$45K of 6 or more people family)
* mental conditions that require other treatment priorities (e.g., suicidal risk, substance abuse, current or past episodes of psychotic disorder, personality disorders)
* medical conditions that severely limit participation, comprehension, or adherence to treatment (e.g., epilepsy, dementia, terminal medical illness) and,
* current usage of antidepressant or mood stabilizers.

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The change of the level of depressive symptoms | From Time 0 (baseline) to Time 1 (at week 8 or 12)
  Measured by the Depression sub-scale of Depression, Anxiety and Stress Scale 21-item version. The subscale has 7 items, each rated from 0 to 3, the total score will be doubled for interpretation of its severity. The higher score indicates the more severe depressive symptoms.
The change of the level of anxiety symptoms | From Time 0 (baseline) to Time 1 (at week 8 or 12)
  Measured by the Anxiety sub-scale of Depression, Anxiety and Stress Scale 21-item version. The subscale has 7 items, each rated from 0 to 3, the total score will be doubled for interpretation of its severity. The higher score indicates the more severe depressive symptoms.
The change of the level of stress symptoms | From Time 0 (baseline) to Time 1 (at week 8 or 12)
  Measured by the Stress sub-scale of Depression, Anxiety and Stress Scale 21-item version. The subscale has 7 items, each rated from 0 to 3, the total score will be doubled for interpretation of its severity. The higher score indicates the more severe depressive symptoms.

SECONDARY OUTCOMES:
The change of subjective quality of life | From Time 0 (baseline) to Time 1 (at week 8 or 12)
  Measured by the Mental Component Summary (MCS) of Short Form 12 version 2. Min: 0, max:100. The higher score indicates better mental health related subjective quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Yu Hai Chen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suen YN, Chen EYH, Wong YC, Ng W, Patwardhan S, Cheung C, Hui CLM, Wong SMY, Wong MTH, Mahtani S. Effects of a culturally adapted counselling service for low-income ethnic minorities experiencing mental distress: a pragmatic randomised clinical trial. BMJ Ment Health. 2023 Aug;26(1):e300788. doi: 10.1136/bmjment-2023-300788. PMID 37597877